CLINICAL TRIAL: NCT05701241
Title: Continuing Somatostatin Analogues Upon Progression in Neuroendocrine Tumour pAtients - The SAUNA Trial
Brief Title: Continuing Somatostatin Analogues Upon Progression in Neuroendocrine Tumour pAtients
Acronym: SAUNA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Erasmus Medical Center (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other); Belgium Health Care Knowledge Centre (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDGE 002337
Record Dates: First submitted 2023-01-05; First posted 2023-01-27 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-04

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumor
Keywords: somatostatin analogues; neuroendocrine tumor
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor; Neuroendocrine Tumors | interventions — Somatostatin; lanreotide; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- somatostatin analogs continuation (Active Comparator): Somatostatin analog (octreotide long-acting release (LAR) 30 mg or lanreotide 120 mg) will be given every four weeks for a duration of 18 months.
  Interventions: Drug: Somatostatin analog
- somatostatin analogs withdrawal (No Intervention): Somatostatin analog treatment (octreotide LAR 30 mg or lanreotide 120 mg) will be withdrawn for a duration of 18 months.

INTERVENTIONS:
Drug: Somatostatin analog — Somatostatin analog treatment every 4 weeks
  Other Names: lanreotide; octreotide; sandostatin; somatuline
  Arms: somatostatin analogs continuation

SUMMARY:
The SAUNA trial is a multi-national, multi-centre, open-label, randomised, controlled, pragmatic clinical trial in patients with advanced, non-functional gastroenteropancreatic (GEP) neuroendocrine tumours (NET) with progressive disease on first-line therapy with somatostatine analogues (SSA). Eligible patients will be divided into two substudies according to the second-line therapy of choice (peptide receptor radionuclide therapy (PRRT) or targeted therapy, at the discretion of the local investigator). Patients within each substudy will be randomised 1:1 between continuation or withdrawal from SSA at the start of second-line systemic therapy. Stratification will occur according to study site and according to the Ki67 value (below 10% (grade 1 and low grade 2) and equal to or above 10% (high grade 2)).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Written informed consent prior to any study-related procedures
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2,
* Histologically-proven diagnosis of locally advanced or metastatic, non-functional, well-differentiated World Health Organisation 2019 grade 1-2 GEP NET
* Documented radiological disease progression on first-line SSA treatment at label dose or higher
* For targeted therapy substudy: indication to start with either sunitinib or everolimus as second-line therapy, according to local investigator
* For PRRT substudy: indication to start with PRRT with Lutetium (177Lu) oxodotreotide as second-line therapy, according to local investigator

Exclusion Criteria:

* Indication for chemotherapy treatment of GEP NET in second-line
* Presence of poorly differentiated grade 3 neuroendocrine carcinoma (NEC), well-differentiated grade 3 NET or rapidly progressive NET
* Prior treatment with everolimus, sunitinib or PRRT
* Contra-indication, proven allergy or other indication than functional NET for the use of a SSA
* Patient showing progressive disease while being on a lower than the registered dose
* Functional NET, defined as the presence of clinical and biochemical evidence of a hormonal NET-related syndrome
* Patient undergoing palliative, systemic oncological treatment for other malignancy than GEP NET
* Concurrent anti-cancer treatment in another investigational trial
* Any abnormal findings at screening, clinical finding, including psychiatric and behavioural problems, or any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might jeopardize the patient's safety or decrease the chance of obtaining satisfactory data needed to achieve the objective(s) of the study
* Pregnant or lactating patient at screening or if the patient wishes to get pregnant during treatment phase of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2023-06-28 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
the difference in progression-free survival (PFS) in patients continuing or stopping second-line therapy with SSAs, as assessed by the blinded local investigator on cross-sectional imaging, according to RECIST 1.1 criteria per substudy | 18 months after start second-line treatment
  PFS
The difference in time to deterioration (TTD) in patients continuing or stopping second-line therapy with SSAs per substudy | 18 months after start second-line treatment
  TTD

SECONDARY OUTCOMES:
progression-free survival rate according to RECIST 1.1 | 18 months after start second-line treatment
  PFS rate
The difference in a pooled progression-free survival of both substudies | 18 months after start second-line treatment
  PFS
The difference in a pooled time to deterioration of both substudies | 18 months after start second-line treatment
  TTD
Overall survival (OS) per substudy and pooled over both substudies | Time until death; assessed up to 5 years after treatment phase
  OS
Overall survival pooled over both substudies | Time until death; assessed up to 5 years after treatment phase
  OS
Response rates (RR) per substudy | 18 months after start second-line treatment
  RR
Response rates over both substudies | 18 months after start second-line treatment
  RR
Quality of life (QoL) measurement with questionnaire | End of study (6.5 years after start second-line treatment)
  QoL measurement with 30-item Quality of Life Questionnaire (QLQ-C30)
Quality of life (QoL) measurement with questionnaire | End of study (6.5 years after start second-line treatment)
  QoL measurement with 21-item QoL questionnaire in the gut, pancreas and liver neuroendocrine tumours (QLQ-GINET21)
Quality of life (QoL) measurement with questionnaire | End of study (6.5 years after start second-line treatment)
  QoL measurement with EuroQol-5 Dimensions-5 Level questionnaire
Cost-effectiveness | End of study (6.5 years after start second-line treatment)
  Health technology assessment (HTA) analysis
Drug safety | 18 months after start second-line treatment
  Safety will be reported in terms of incidence and severity of (serious) adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Marc Peeters, MD, Principal Investigator — University Hospital, Antwerp
Locations (19):
- Belgium (13):
  - AZ Klina, Brasschaat, Antwerp
  - AZ Rivierenland, Rumst, Antwerp
  - Ghent University Hospital, Ghent, East Flanders
  - VITAZ, Sint-Niklaas, East-Flanders
  - University Hospital Leuven, Leuven, Flemish Brabant
  - Grand Hôpital de Charleroi, Charleroi, Hainaut
  - AZ Monica, Antwerp
  - GZA, Antwerp
  - Ziekenhuis Netwerk Antwerpen, Antwerp
  - Cliniques Universitaires Saint-Luc, Brussels
  - H.U.B., Brussels
  - Antwerp University Hospital, Edegem
  - Centre Hospitalier Universitaire Sart Tilman, Liège
- Netherlands (6):
  - Rijnstate, Arnhem, Gelderland
  - Maastricht UMC+, Maastricht, Limburg
  - Maxima Medisch Centrum, Eindhoven, North Brabant
  - Amsterdam UMC, Amsterdam, North Holland
  - UMC Groningen, Groningen
  - Erasmus MC, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chhajlani S, Kuiper J, Beutels P, Borbath I, Dercksen W, Deroose CM, Heemskerk S, Polinder S, Roelant E, Smits E, Verhaegen I, Van der Massen I, Walenkamp A, de Herder WW, Peeters M, Hofland J, Vandamme T; SAUNA investigators and the Dutch Belgian Neuroendocrine Tumor Society (DBNETS). Somatostatin analogue continuation upon progression in patients with gastroenteropancreatic neuroendocrine tumour (SAUNA trial): a randomised controlled trial protocol. BMJ Open. 2025 Jul 3;15(7):e099996. doi: 10.1136/bmjopen-2025-099996. PMID 40615151